CLINICAL TRIAL: NCT06350760
Title: Transdiagnostic, Indicated Preventive Intervention for Adolescents At High Risk of Emotional Problems With Add-On Modules (PROCARE-I+)
Brief Title: Transdiagnostic, Indicated Preventive Intervention for Adolescents At High Risk of Emotional Problems W/Add-On Modules
Acronym: PROCARE-I+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other); University Rovira i Virgili (Other); University of Miami (Other)
Responsible Party: Principal Investigator, LuisJoaquin Garcia-Lopez, Full Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UJA_PROCARE-I+
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Disorders and Symptoms; Depressive Symptoms
Keywords: transdiagnostic; emotional disorders; anxiety; depression; adolescents; child and youth population; indicated prevention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: To-arm interventions are carried out, measuring at the pre-intervention moment and at the post-intervention moment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PROCARE-I (UP-A for indicated purposes) (Experimental): To ensure cost-effectiveness, PROCARE-I intervention will be designed as a brief 8-session child-focused programme by adapting the core modules from UP-A, along with one individual session with adolescent and parents. Sessions will be delivered in reduced groups, using a typical indicated preventive intervention format focused on cost-effectiveness.
  Interventions: Behavioral: Active control condition
- PROCARE-I+ 8-session (for indicated purposes) (Experimental): PROCARE-I+ intervention will be designed as a brief 8-session with 4 additonal sessions (add-on modules) child-focused programme by adapting the core modules from UP-A. Sessions will be delivered in reduced groups, using a typical indicated preventive intervention format focused on cost-effectiveness.
  Interventions: Behavioral: PROCARE-I+ 8-session

INTERVENTIONS:
Behavioral: Active control condition — The active control condition will be based on PROCARE protocol, which was put into practice in PROCARE-I, in 2021.
  Arms: PROCARE-I (UP-A for indicated purposes)
Behavioral: PROCARE-I+ 8-session — The active control condition will be based on PROCARE protocol, which was put into practice in PROCARE-I, in 2021. In addition, PROCARE-I+ adds additional modules, which allow adolescents to be provided with tools to address the risk factors they present.
  Arms: PROCARE-I+ 8-session (for indicated purposes)

SUMMARY:
PROCARE is a preventive intervention that has shown its effectiveness in selective prevention to reduce young people's risk of developing emotional problems. In this study, an uncontrolled pre-post study is carried out where this personalized transdiagnostic preventive intervention in online mode is applied in the indicated population, with the following objectives: 1) provide data about whether there are improvements in the emotional state of adolescents after implementing PROCARE-I+; and 2) evaluate if there is any risk factor that predicts anxiety-depressive symptoms and/or emotional difficulties. The sample was made up of 30 adolescents who showed symptoms of anxiety and/or depression and a high risk of developing an emotional disorder and who benefited from the preventive, transdiagnostic, online and personalized intervention called PROCARE-I+. After the analysis of the data collected at the pre-intervention and post-intervention time, the data revealed that the intervention had an impact on improving the emotional state of the adolescents in terms of anxious-depressive symptomatology, quality of life and emotional regulation. On the other hand, the data revealed the absence of predictive relationships between the presence of a risk factor and suffering from symptoms of anxiety and depression; In contrast, predictive relationships were found between the presence of the family risk factor and suffering from some emotional difficulty.

DETAILED DESCRIPTION:
The general objetive of PROCARE-I+ is to implement and evaluate an indicated 8-session preventive group intervention with add-on modules for adolescents aged 12-18 at high risk of emotional disorders like anxiety and depression. The intervention will be based on the Unified protocol for transdiagnostic treatment of emotional disorders in adolescents (UP-A), already proven as effective in the US, but adapted with indicated prevention purposes in Spain thanks support of main author of the protocol (Prf. Ehrenreich-May). It will be culturally-adapted and designed to be an acceptable, scalable, and sustainable indicated prevention program.

METHODOLOGY: In order to achieve this objetive, PROCARE-I+ working plan will be divided into 3 steps. Firstly, in order to identify adolescents at high risk of suffering emotional disorders (anxiety and depression), the following self-reports will be administered to adolescents: Strengths and Difficulties Questionnaire (SDQ) to evaluate adolescents at-risk of emotional disorders, and the Revised Child Anxiety and Depression Scale-30 (RCADS-30) will screen for presence/absence of emotional symptomatology. Then, ADIS5-C/P will be administered to rule-out presence of anxiety and/or mood disorders. Valuing voices from stakeholders and end-users, the investigators will focus on the study of the influence of the above described variables. Third, the investigators will test PROCARE-I with add-on modules.

IMPACT: The following study will be taken as a pilot study that will allow us to know the strengths and weaknesses of PROCARE-I with add-on modules in order to make future improvements.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from adolescent and legal guardian
* able to attend prevention modules on his/her own
* language competence
* Strengths and Difficulties Questionnaire ""probable diagnoses"
* score above cut-off for Revised Child Anxiety and Depression Scale-30
* having incipient symptoms on an emotional level in ADIS 5 C/P
* absence of anxiety and/or mood disorders

Exclusion Criteria:

* in- or outpatient
* concomitant psychological/psychiatric treatment
* acute suicidality
* general medical contraindications that hamper attendance to prevention modules
* have been diagnosed with a neurodevelopmental disorder
* Strengths and Difficulties Questionnaire "unlikely" or "possible diagnoses"
* presence of mood and/or anxiety disorders

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported anxiety and mood symptomatology | Baseline to 7 months after start of interventions
  The study's primary outcome was self-reported anxiety and mood symptomatology as assessed by Revised Child Anxiety Depression Scale (RCADS-30). Total scores range from 0 to 90. Higher scores mean a worse outcome
Factors associated with adolescents' mental health | Baseline to 7 months after start of interventions
  The study's primary outcome was self-reported risk and protective factors level of emotional disorders as assessed by Strengths and Difficulties Questionnaire (SDQ). Total scores range from 0 to 50. Higher scores mean a worse outcome.
Resilience measure | Baseline to 7 months after start of interventions
  This primary measure was intended to measure the resilience of adolescents through 10 items with 5 response options. Scores range from 0 to 40. The higher the score, the greater the resilience.
Health-related quality of life | Baseline to 7 months after start of interventions
  Secondary outcome assessed included self-reported changes in health-related quality of life as assessed by KIDSCREEN-10. Total scores range from 10 to 50. Higher scores mean a better outcome.
Absence of emotional disorders | Baseline to 7 months after start of interventions
  The study's primary outcome was absence of any emotional disorders over the long-term measured by the ADIS-5-C/P

SECONDARY OUTCOMES:
Economic evaluations | Baseline to 7 months after start of interventions
  Implementation service costs (training, program materials, provider salaries), costs to school system, and later health costs saved for preventing emotional problems that could narrow cumulative disparities in mental health and disadvantage later in life.
Psychological flexibility | Baseline to 7 months after start of interventions
  Psychological flexibility as assessed by Willingness and Action Measure for Children and Adolescents (WAM-C/A).
  Total scores range from 0 to 56. Higher scores mean a better outcome.
Emotional regulation | Baseline to 7 months after start of interventions
  The Difficulties in Emotion Regulation Scale (DERS). Scores range from 0 to 150. The higher the score, the greater the difficulties in emotional regulation.

OTHER OUTCOMES:
Bullying | Baseline to 7 months after start of interventions
  Cyberbullying. peer bullying screening. Scores range from 0 to 40. The higher the score, the greater the role played in bullying (aggressor, victim, observer).
Expressed Emotion | Baseline to 7 months after start of interventions
  Expressed Emotion Evaluation Questionnaire. The scores range from 1 to 7. The higher the score, the greater the difficulties in the family communication style.
Ecoanxiety | Baseline to 7 months after start of interventions
  Climate Anxiety Scale. Scores range from 13 to 52. The higher the score, the greater the climate anxiety.
Exam anxiety | Baseline to 7 months after start of interventions
  Test anxiety questionnaire adapted for ESO and Baccalaureate. Scores range from 35 to 140. The higher the score, the greater the anxiety before the exams.
Videogames addiction | Baseline to 7 months after start of interventions
  Game Addiction Scale for Adolescents (GASA). Scores range from 0 to 28. The higher the score, the greater the risk of video game addiction.
Smartphone addiction | Baseline to 7 months after start of interventions
  Smartphone Addiction Scale - Short Version (SAS-SV). Scores range from 10 to 70. The higher the score, the greater the risk of smartphone addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Joaquín García-López, Ph. D., Principal Investigator — University of Jaén
Locations (3):
- Spain (3):
  - Universidad Miguel Hernández, Elche, Alicante
  - University of Jaén, Jaén, Jaen
  - Universitat Rovira i Virgili, Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: Yes
Authors of secondary analyses using shared data will attest that their use was in accordance with the terms (if any) agreed to upon their receipt. They will also reference the source of the data using its unique, persistent identifier to provide appropriate credit to those who generated it and allow searching for the studies it has supported. Authors of secondary analyses will explain completely how theirs differ from previous analyses. In addition, those who generate and then share clinical trial data will deserve substantial credit for their efforts. Those using data collected by others will seek collaboration with those who collected the data. As collaboration will not always be possible, practical, or desired, the efforts of those who generated the data will be recognized.
Supporting Information: CSR
Time Frame: From June 2024
Access Criteria: upon request to authors

REFERENCES:
- [Background] Ehrenreich-May, J.; & Kennedy, S.M. (2022). Protocolo unificado para el tratamiento transdiagnóstico de los trastornos emocionales en niños y adolescentes: Manual del terapeuta. Ediciones Pirámide.
- [Background] Vivas-Fernandez M, Garcia-Lopez LJ, Piqueras JA, Muela-Martinez JA, Canals-Sans J, Espinosa-Fernandez L, Jimenez-Vazquez D, Diaz-Castela MDM, Morales-Hidalgo P, Rivera M, Ehrenreich-May J. Randomized controlled trial for selective preventive transdiagnostic intervention for adolescents at risk for emotional disorders. Child Adolesc Psychiatry Ment Health. 2023 Jan 12;17(1):7. doi: 10.1186/s13034-022-00550-2. PMID 36635735